CLINICAL TRIAL: NCT02479373
Title: "Joint Fitness": A Double-Armed Controlled Intervention to Assess the Safety and Effectiveness of Resistance Exercise Training on Muscle, Bone, Strength, Symptoms, Quality of Life and Biological Parameters in Children and Young Adults With JIA
Brief Title: Exercise and Body Composition in Juvenile Idiopathic Arthritis
Acronym: Joint Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: NA00071505; 5R21AR062269-02 (NIH)
Record Dates: First submitted 2015-05-01; First posted 2015-06-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Arthritis, Juvenile
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: Control and participant groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise (RE) (Experimental): Those assigned to RE will complete baseline and post-testing assessments and participate in 12 weeks of individually-supervised resistance exercise, which will take place in the exercise facility on the Johns Hopkins Bayview Medical Center Campus. Exercises will be performed on Ren-Ex Machines. This equipment is suitable for the proposed study because it provides ultra-low friction movement which creates a personalized resistance profile, which minimizes force on joints and thereby reduces the risk of joint trauma and injury.
  Interventions: Other: Ren-Ex Machine; Other: Dual-Emission X-ray Absorptiometry (DEXA) scan; Other: Biodex dynamometer; Other: Sub-maximal test; Other: Quality of life questionnaires
- Control Group (CG) (Other): Those assigned to the CG will complete baseline and post-testing assessments and will also be given JIA educational materials, including physical activity and exercise recommendations from the American Academy of Pediatrics (AAP) Council on Sports Medicine and Fitness (COSMF).
  Interventions: Other: Dual-Emission X-ray Absorptiometry (DEXA) scan; Other: Biodex dynamometer; Other: Sub-maximal test; Other: Quality of life questionnaires

INTERVENTIONS:
Other: Ren-Ex Machine — The exercise is performed once per week with individualized instruction using moderate resistance on Ren-Ex Machines, ultra-low-friction equipment to minimize force on joints.
  Arms: Resistance Exercise (RE)
Other: Dual-Emission X-ray Absorptiometry (DEXA) scan — To study body composition
Other: Biodex dynamometer — To study muscle strength
  Other Names: Isokinetic strength testing
Other: Sub-maximal test — To study lung capacity, a sub-maximal (limited exercise) test on a stationary bicycle is performed.
Other: Quality of life questionnaires

SUMMARY:
This research is being done to see if resistance exercise (RE) is safe and has a positive effect on children and young adults with juvenile idiopathic arthritis (JIA).

JIA is an inflammatory autoimmune disease that can cause severe impairment and disability. JIA can cause bone loss and decreased muscle strength. The medications used to treat JIA can also have negative effects on growth and development, strength, and ability to function. RE is performing movements in a slow and controlled fashion (i.e., no speeding up or using force in the lifting and lowering of the weight) to lessen force on the joints and tissues. This study will be using Ren-Ex exercise equipment to perform RE.

Currently the American College of Rheumatology recommends exercise for patients with arthritis. This exercise includes range of motion exercise to protect joint mobility as well as low resistance and aerobic exercise (AE) to protect muscle mass, bone health, and fitness. However, a recent study showed no major differences in functionality or quality of life between patients who performed AE and those who did not perform AE. There is a need for more data on the impact of RE on children with JIA. Children and young adults aged 10 to 21 with juvenile idiopathic arthritis may join.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology criteria for polyarticular JIA
* Stable medical therapy

Exclusion Criteria:

* Non-English speaking
* Pregnancy
* Currently breast feeding
* Cognitive impairment as determined by PI (patient is not responsible for making their own health care decisions)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Total Body Dual-Emission X-ray Absorptiometry (DEXA) Scan | Baseline and 12 weeks
  Total and lean body mass and fat mass will be determined
Change in BMI | Baseline and 12 weeks
Change in Lower and upper extremity strength testing | Baseline and 12 weeks
  Isokinetic strength testing with a Biodex dynamometer to measure peak torque

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline and 12 weeks
Change in Erythrocyte sedimentation rate (ESR) | Baseline and 12 weeks
Change in Quality of Life | Baseline and 12 weeks
  Questionnaire administration
Change in C-reactive protein (CRP) | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sule, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No